CLINICAL TRIAL: NCT03480243
Title: An Open-label, Fixed-sequence Study in Healthy Study Participants to Evaluate the Effect of Coadministered Erythromycin on the Pharmacokinetics and Safety of Padsevonil
Brief Title: Study to Evaluate the Effect of Coadministered Erythromycin on the Pharmacokinetics and Safety of Padsevonil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: UP0057; 2017-004694-13 (EudraCT Number)
Record Dates: First submitted 2018-03-21; First posted 2018-03-29 (Actual); Results first posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Pharmacokinetics
Keywords: Padsevonil
MeSH Terms: interventions — padsevonil; Erythromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Padsevonil and Erythromycin (Experimental): Treatment Period 1 (Day 1 to Day 11):
  * Padsevonil 100 mg twice daily (bid) on Day 1 to Day 4
  * Padsevonil 100 mg single dose on Day 5
  * 1 week of wash-out (from evening of Day 5 to Day 11)
  Treatment Period 2 (Day 12 to 22):
  * Padsevonil 100 mg twice daily (bid) on Day 12 to Day 15
  * Padsevonil 100 mg single dose on Day 16
  * 1 week of wash-out (from evening of Day 16 to Day 22)
  Treatment Period 3 (Day 23 to Day 38):
  * Erythromycin 500 mg twice daily (bid) on Day 23 to Day 25
  * Padsevonil 100 mg bid and erythromycin 500 mg bid on Day 26 to Day 32
  * Padsevonil 100 mg single dose on Day 33
  * Erythromycin 500 mg twice daily (bid) on Day 33 to Day 36
  * Erythromycin 500 mg single dose on Day 37
  Interventions: Drug: Padsevonil (UCB0942); Drug: Erythromycin

INTERVENTIONS:
Drug: Padsevonil (UCB0942) — * Pharmaceutical Form: film-coated tablet
  * Route of Administration: Oral use
Drug: Erythromycin — * Pharmaceutical Form: film-coated tablet
  * Route of Administration: Oral use

SUMMARY:
The purpose of this study is to evaluate and compare the Pharmacokinetics (PK) of concomitant administration of Padsevonil (PSL) in the presence and absence of erythromycin in healthy study participants.

ELIGIBILITY:
Inclusion Criteria:

* Study participant is male or female and between 18 and 55 years of age (inclusive)
* Study participant is of a body weight of at least 50 kg for males and 45 kg for females, as determined by a body mass index (BMI) between 18 and 30 kg/m^2
* Female study participants use an efficient form of contraception for the duration of the study (unless menopausal). Hormonal contraception may be susceptible to an interaction with the Investigational Medicinal Product (IMP), which may reduce the efficacy of the contraception method. The potential for reduced efficacy of any hormonal contraception methods requires that a barrier method (preferably male condom) also be used
* Study participant has clinical laboratory test results within the local reference ranges or values are considered as not clinically relevant by the investigator and approved by the UCB Study Physician
* Study participant has Blood Pressure (BP) and pulse rate within normal range in supine position after 10 minutes of rest
* Male study participant agrees that, during the study period, when having sexual intercourse with a woman of childbearing potential, he will use an efficient barrier contraceptive (condom plus spermicide) AND that the respective partner will use an additional efficient contraceptive method

Exclusion Criteria:

* Study participant has previously received Investigational Medicinal Product (IMP) in this study
* Study participant has participated in another study of an IMP (or a medical device) within the previous 3 months before Screening (or within 5 half-lives for the IMP, whichever is longer) or is currently participating in another study of an IMP (or a medical device)
* Study participant has a history of drug or alcohol dependency within the previous 6 months or tests positive for alcohol (breath test) and/or drugs of abuse (urine test) at the Screening Visit or at any time during confinement
* Study participant has made a blood or plasma donation or has had a comparable blood loss (>400 mL) within the last 3 months prior to the Screening Visit
* Study participant smokes more than 5 cigarettes per day (or equivalent) or has done so within 6 months prior to the Screening Visit
* Study participant is taking any concomitant medication currently or within 2 weeks prior to the first day of dosing with the exception of paracetamol (acetaminophen)
* Study participant has any clinically relevant Electrocardiogram (ECG) finding at the Screening Visit or confinement
* Study participant has a history within the last 5 years or present condition of malignancy, with the exception of basal cell carcinoma
* Female study participant tests positive for pregnancy, plans to get pregnant during the participation in the study, or who is breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0057 001, London, United Kingdom

REFERENCES:
- [Derived] Chanteux H, MacPherson M, Kramer H, Otoul C, Okagaki T, Rospo C, De Bruyn S, Watling M, Bani M, Sciberras D. Overview of preclinical and clinical studies investigating pharmacokinetics and drug-drug interactions of padsevonil. Expert Opin Drug Metab Toxicol. 2024 Aug;20(8):841-855. doi: 10.1080/17425255.2024.2373108. Epub 2024 Jul 9. PMID 38932723

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in March 2018 and concluded in August 2018.
Pre-assignment Details: Participant Flow refers to the Full Analysis Set (FAS).
Groups:
- Padsevonil and/or Erythromycin: The study participants received treatment as follows:
  Treatment Period 1: From Day 1 to Day 11:
  * Padsevonil 100 mg twice daily (bid) on Day 1 to Day 4
  * Padsevonil 100 mg single dose on Day 5
  * 1 week of wash-out (from evening of Day 5 to Day 11).
  Treatment Period 2: From Day 12 to Day 22:
  * Padsevonil 100 mg bid on Day 12 to Day 15
  * Padsevonil 100 mg single dose on Day 16
  * 1 week of wash-out (from evening of Day 16 to Day 22).
  Treatment Period 3: From Day 23 to 37
  Treatment Period 3a:
  -Erythromycin 500 mg bid on Day 23 to Day 25.
  Treatment Period 3b:
  * Padsevonil 100 mg bid and erythromycin 500 mg bid on Day 26 to Day 32
  * Padsevonil 100 mg single dose on Day 33
  * Erythromycin 500 mg bid on Day 33.
  Treatment Period 3c:
  - Erythromycin 500 mg bid on Day 34 to Day 37.
Period: Padsevonil (Period 1)
Arm/Group | Padsevonil and/or Erythromycin
Started | 28
Completed | 28
Not Completed | 0
Period: Padsevonil (Period 2)
Arm/Group | Padsevonil and/or Erythromycin
Started | 28
Completed | 27
Not Completed | 1
Not completed — Consent withdrawal by subject | 1
Period: Erythromycin (Period 3a)
Arm/Group | Padsevonil and/or Erythromycin
Started | 27
Completed | 27
Not Completed | 0
Period: Padsevonil and Erythromycin (Period 3b)
Arm/Group | Padsevonil and/or Erythromycin
Started | 27
Completed | 26
Not Completed | 1
Not completed — Un-cooperative behaviour | 1
Period: Erythromycin (Period 3c)
Arm/Group | Padsevonil and/or Erythromycin
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Full Analysis Set (FAS) which consisted of all study participants who have signed the Informed Consent Form (ICF) and received the investigational medicinal product (IMP).
Arm/Group | Padsevonil and/or Erythromycin
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black | 1
  White | 24
  Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Padsevonil for Single Dose
Description: Cmax: The maximum observed plasma concentration of padsevonil for single dose . Cmax was expressed in nanograms per milliliter (ng/mL).
Time Frame: Predose and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose on Day 1, 12, and 26
Population: The Pharmacokinetic Per-Protocol Set (PK-PPS) was a subset of the FAS, consisting of those study participants who had no important protocol deviations affecting the PK parameters and for whom a sufficient number of samples were available to determine at least 1 PK parameter. As per the planned analysis, data was summarized by treatment periods.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Padsevonil (Period 1) (PK-PPS): The study participants, of a single cohort, received Padsevonil during the Treatment Period 1 as follows: From Day 1 to Day 11:
  * Padsevonil 100 mg bid on Day 1 to Day 4
  * Padsevonil 100 mg single dose on Day 5
  * 1 week of wash-out (from evening of Day 5 to Day 11). Study participants formed the Pharmacokinetic-Per Protocol Set (PK-PPS).
- Padsevonil (Period 2) (PK-PPS): The study participants, of a single cohort, received Padsevonil during the Treatment Period 2 as follows: From Day 12 to Day 22:
  * Padsevonil 100 mg bid on Day 12 to Day 15
  * Padsevonil 100 mg single dose on Day 16
  * 1 week of wash-out (from evening of Day 16 to Day 22). Study participants formed the PK-PPS.
- Padsevonil and Erythromycin (Period 3b) (PK-PPS): The study participants, of a single cohort, received Padsevonil and Erythromycin during the second part of the Treatment Period 3b as follows:
  * Padsevonil 100 mg bid and erythromycin 500 mg bid on Day 26 to Day 32
  * Padsevonil 100 mg single dose on Day 33
  * Erythromycin 500 mg bid on Day 33. Study participants formed the PK-PPS.
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 27
ng/mL | 366.6 (38.8) | 385.3 (40.9) | 697.4 (46.9)
Statistical Analysis 1: Comparison: Padsevonil (Period 1) (PK-PPS) vs Padsevonil and Erythromycin (Period 3b) (PK-PPS); The analysis of variance model included the fixed effects period (1, 2 or 3b) and participant as a random effect; Test type: Other; ANOVA; Cmax Estimate Ratio = 1.90, 90% CI 2-sided [1.59 to 2.27]
Statistical Analysis 2: Comparison: Padsevonil (Period 2) (PK-PPS) vs Padsevonil and Erythromycin (Period 3b) (PK-PPS); The analysis of variance model included the fixed effects period (1, 2 or 3b) and participant as a random effect; Test type: Other; ANOVA; Cmax Estimate Ratio = 1.81, 90% CI 2-sided [1.51 to 2.16]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 12 Hours (AUC(0-12)) of Padsevonil for Single Dose
Description: AUC(0-12): The area under the plasma concentration-time curve from time zero to 12 hours of padsevonil for single dose . AUC(0-12) was expressed in hours times nanograms per milliliter (hours*ng/mL).
Time Frame: Predose and 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, and 12 hours postdose on Day 1, 12, and 26
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 27
hours*ng/mL | 1428 (40.7) | 1571 (41.8) | 2576 (47.0)
Statistical Analysis 1: Comparison: Padsevonil (Period 1) (PK-PPS) vs Padsevonil and Erythromycin (Period 3b) (PK-PPS); The analysis of variance model included the fixed effects period (1, 2 or 3b) and participant as a random effect; Test type: Other; ANOVA; AUC Estimate Ratio = 1.80, 90% CI 2-sided [1.50 to 2.17]
Statistical Analysis 2: Comparison: Padsevonil (Period 2) (PK-PPS) vs Padsevonil and Erythromycin (Period 3b) (PK-PPS); The analysis of variance model included the fixed effects period (1, 2 or 3b) and participant as a random effect; Test type: Other; ANOVA; AUC Estimate Ratio = 1.64, 90% CI 2-sided [1.36 to 1.97]

3. Primary Outcome: Maximum Observed Steady-state Plasma Concentration (Cmax, ss) of Padsevonil for Multiple Doses
Description: Cmax, ss: The maximum observed steady-state plasma concentration of padsevonil for multiple doses. Cmax, ss was expressed in nanograms per millilitre (ng/mL).
Time Frame: Blood samples were taken at specific time points from pre-dose to 72 hours post last dose of Padsevonil (PSL) (Treatment Period 1 and 2); from pre-dose to 120 hours post last dose of PSL (Treatment Period 3)
Population: The Pharmacokinetic Per-Protocol Set (PK-PPS) was a subset of the FAS, consisting of those study participants who had no important protocol deviations affecting the PK parameters and for whom a sufficient number of samples were available to determine at least 1 PK parameter. As per the planned analysis, data was summarized by treatment periods. Here, number of participants were included who were evaluable for the assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 26
ng/mL | 475.0 (38.4) | 473.9 (43.7) | 1010 (45.7)
Statistical Analysis 1: Comparison: Padsevonil (Period 1) (PK-PPS) vs Padsevonil and Erythromycin (Period 3b) (PK-PPS); The analysis of variance model included the fixed effects period (1, 2 or 3b) and participant as a random effect; Test type: Other; ANOVA; Cmax,ss Estimate Ratio = 2.13, 90% CI 2-sided [1.77 to 2.55]
Statistical Analysis 2: Comparison: Padsevonil (Period 2) (PK-PPS) vs Padsevonil and Erythromycin (Period 3b) (PK-PPS); The analysis of variance model included the fixed effects period (1, 2 or 3b) and participant as a random effect; Test type: Other; ANOVA; Cmax,ss Estimate Ratio = 2.13, 90% CI 2-sided [1.78 to 2.56]

4. Primary Outcome: Area Under the Plasma Concentration-time Curve Over a Dosing Interval (12 Hours) (AUCtau) of Padsevonil for Multiple Doses
Description: AUCtau: The area under the plasma concentration-time curve over a dosing interval (12 hours) of padsevonil for multiple doses. AUC(tau) was expressed in hours times nanograms per millilitre (hours*ng/mL).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 26
hours*ng/mL | 2049 (41.1) | 2274 (47.1) | 5073 (55.9)
Statistical Analysis 1: Comparison: Padsevonil (Period 1) (PK-PPS) vs Padsevonil and Erythromycin (Period 3b) (PK-PPS); The analysis of variance model included the fixed effects period (1, 2 or 3b) and participant as a random effect; Test type: Other; ANOVA; AUCtau Estimate Ratio = 2.48, 90% CI 2-sided [2.02 to 3.03]
Statistical Analysis 2: Comparison: Padsevonil (Period 2) (PK-PPS) vs Padsevonil and Erythromycin (Period 3b) (PK-PPS); The analysis of variance model included the fixed effects period (1, 2 or 3b) and participant as a random effect; Test type: Other; ANOVA; AUCtau Estimate Ratio = 2.23, 90% CI 2-sided [1.82 to 2.73]

5. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Padsevonil for Single Dose
Description: Tmax: The time of maximum plasma concentration of padsevonil for single dose. Tmax was expressed in hours (h).
Time Frame: Blood samples were taken at specific time points from pre-dose to 12 hours post first dose of Padsevonil for each Treatment Period
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 27
hours | 3.000 [1.00 to 4.05] | 1.500 [0.500 to 4.00] | 1.500 [0.750 to 3.02]

6. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of Padsevonil for Single Dose
Description: Cmin: The minimum observed plasma concentration of padsevonil for single dose. Cmin was expressed in nanograms per millilitre (ng/mL).
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 27
ng/mL | 2.857 (100.9) | 5.643 (147.8) | 4.286 (172.5)

7. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of Padsevonil for Multiple Doses
Description: Tmax: The time of maximum plasma concentration of padsevonil for multiple doses. Tmax was expressed in hours (h).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 26
hours | 1.750 [0.500 to 4.00] | 1.500 [0.500 to 4.00] | 2.000 [0.750 to 4.00]

8. Secondary Outcome: Apparent Terminal Elimination Half-life at Steady-state (t1/2,ss) of Padsevonil for Multiple Doses in Plasma
Description: t½,ss: The apparent terminal elimination half-life at steady-state of padsevonil for multiple doses in plasma. t1/2, ss was expressed in hours (h).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Median (Full Range); unit: hours
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 26
hours | 6.465 [4.44 to 11.0] | 6.649 [2.04 to 14.3] | 8.548 [5.54 to 26.9]

9. Secondary Outcome: Predose Observed Plasma Concentration (Ctrough) of Padsevonil for Multiple Doses
Description: Ctrough: The predose observed plasma concentration of padsevonil for multiple doses. Ctrough was expressed in nanograms per millilitre (ng/mL).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 26
ng/mL | 57.03 (69.0) | 68.57 (85.1) | 182.6 (95.5)

10. Secondary Outcome: Apparent Total Clearance at Steady-state (CL/Fss) of Padsevonil for Multiple Doses in Plasma
Description: CL/Fss: The apparent total clearance at steady-state of padsevonil for multiple doses in plasma. CL/Fss was expressed in milliliters per hour (mL/hour).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hour
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 26
mL/hour | 48810 (41.1) | 43970 (47.1) | 19710 (55.9)

11. Secondary Outcome: Apparent Elimination Rate Constant (Lambdaz) of Padsevonil for Multiple Doses in Plasma
Description: lambdaz: The apparent elimination rate constant of padsevonil for multiple doses in plasma. Lambdaz was expressed in liters per hour (l/hour).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: l\hour
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 26
l\hour | 0.1049 (27.9) | 0.1006 (36.2) | 0.07975 (34.5)

12. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Padsevonil Metabolites (1 and 2) for Single Dose
Description: Cmax: The maximum plasma concentration of padsevonil metabolites (1 and 2) for single dose. Cmax was expressed in nanograms per milliliter (ng/mL).
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 27
ng/mL
  Metabolite 1 | 166.6 (29.1) | 158.7 (34.5) | 189.5 (29.8)
  Metabolite 2 | 110.5 (33.4) | 94.47 (44.2) | 108.3 (49.6)

13. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to 12 Hours (AUC(0-12)) of Padsevonil Metabolites (1 and 2) for Single Dose
Description: AUC(0-12): The area under the plasma concentration-time curve from time zero to 12 hours of padsevonil metabolites (1 and 2) for single dose. AUC(0-12) was expressed in hours times nanograms per milliliter (hours*ng/mL).
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 27
hours*ng/mL
  Metabolite 1 | 828.3 (24.2) | 824.3 (25.5) | 905.6 (29.7)
  Metabolite 2 | 596.5 (39.0) | 534.4 (43.9) | 599.5 (49.5)

14. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over a Dosing Interval (12 Hours) (AUCtau) of Padsevonil Metabolites (1 and 2) for Multiple Doses
Description: AUCtau: The area under the plasma concentration-time curve over a dosing interval (12 hours) of padsevonil metabolites (1 and 2) for multiple doses. AUCtau was expressed in hours times nanograms per milliliter (hours*ng/mL).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*ng/mL
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 26
hours*ng/mL
  Metabolite 1 | 1748 (35.1) | 1993 (40.8) | 2625 (46.1)
  Metabolite 2 | 775.1 (37.4) | 813.1 (40.5) | 799.0 (38.5)

15. Secondary Outcome: Maximum Observed Steady-state Plasma Concentration (Cmax, ss) of Padsevonil Metabolites (1 and 2) for Multiple Doses
Description: Cmax, ss: The maximum observed steady-state plasma concentration of padsevonil metabolites (1 and 2) for multiple doses. Cmax, ss was expressed in nanograms per millilitre (ng/mL).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 26
ng/mL
  Metabolite 1 | 232.3 (27.1) | 258.3 (32.3) | 310.3 (46.0)
  Metabolite 2 | 118.6 (29.3) | 113.3 (36.8) | 101.8 (37.1)

16. Secondary Outcome: Metabolite-to-parent Ratio for Cmax of Padsevonil Metabolites (1 and 2) in Plasma
Description: Metabolite-to-parent ratio calculated as: Cmax of padsevonil metabolites (1 and 2) divided by Cmax of padsevonil following a single dose in plasma. Metabolite-to-parent ratio for Cmax was expressed as ratio.
Time Frame: Blood samples were taken at specific time points from pre-dose to 12 hours post dose of Padsevonil for each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 27
ratio
  Metabolite 1 | 0.4544 (40.6) | 0.4119 (45.5) | 0.2717 (49.5)
  Metabolite 2 | 0.3015 (66.8) | 0.2452 (77.1) | 0.1552 (94.3)

17. Secondary Outcome: Metabolite-to-parent Ratio for AUC(0-12) of Padsevonil Metabolites (1 and 2) in Plasma
Description: Metabolite-to-parent ratio calculated as: AUC(0-12)of padsevonil metabolites (1 and 2) divided by AUC(0-12) of padsevonil following a single dose in plasma. Metabolite-to-parent ratio for AUC(0-12) was expressed as ratio.
Time Frame: as for outcome 5
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 27
ratio
  Metabolite 1 | 0.5799 (39.7) | 0.5246 (42.8) | 0.3515 (48.9)
  Metabolite 2 | 0.4176 (70.0) | 0.3401 (78.7) | 0.2327 (97.1)

18. Secondary Outcome: Metabolite-to-parent Ratio for AUCtau of Padsevonil Metabolites (1 and 2) in Plasma
Description: Metabolite-to-parent ratio calculated as: AUCtau of padsevonil metabolites (1 and 2) divided by AUCtau of padsevonil following multiple dosing in plasma. Metabolite-to-parent ratio for AUCtau was expressed as ratio.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 26
ratio
  Metabolite 1 | 0.8533 (34.9) | 0.8766 (38.7) | 0.5174 (48.2)
  Metabolite 2 | 0.3783 (63.4) | 0.3576 (75.5) | 0.1575 (88.5)

19. Secondary Outcome: Renal Clearance (CLr) of Padsevonil and Metabolites (1 and 2) for Single Dose in Urine
Description: CLr: The renal clearance of padsevonil and its metabolites (1 and 2) for single dose in urine. CLr was expressed in milliliters per hour (mL/hour).
Time Frame: Urine samples were taken 0 to 12 hours post first dose of Padsevonil during each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hour
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 27
mL/hour
  Padsevonil | 27.40 (54.3) | 25.80 (73.0) | 19.36 (60.2)
  Metabolite 1 | 253.7 (47.8) | 283.0 (60.1) | 255.0 (53.9)
  Metabolite 2 | 17640 (19.6) | 17630 (21.2) | 16290 (20.7)

20. Secondary Outcome: Renal Clearance (CLr) of Padsevonil and Metabolites (1 and 2) for Multiple Doses in Urine
Description: CLr: The renal clearance of padsevonil and its metabolites (1 and 2) for multiple doses in urine. CLr was expressed in milliliters per hour (mL/hour).
Time Frame: Urine samples were taken 0 to 12 hours, 12 to 24 hours,and 24 to 48 hours post last PSL dose during Treatment Period 1 and 2; 0 to 12 hours, 12 to 24 hours, 24 to 48 hours, 48 to 72 hours, and 72 to 96 hours post last dose of PSL during Treatment Period 3
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hours
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 26
mL/hours
  Padsevonil | 28.43 (58.0) | 25.24 (59.7) | 25.12 (56.1)
  Metabolite 1 | 335.0 (50.2) | 325.4 (40.8) | 311.4 (51.7)
  Metabolite 2 | 19390 (24.9) | 18530 (20.7) | 16470 (27.6)

21. Secondary Outcome: Cumulative Amount (Ae) of Padsevonil and Metabolites (1, 2, and 3) Excreted Into the Urine for Single Dose
Description: Ae: The cumulative amount of padsevonil and its metabolites (1, 2, and 3) excreted into the urine for single dose. Ae was expressed in milligrams (mg).
Time Frame: Urine samples were taken 0 to 12 hours post first dose of Padsevonil during each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 27
milligrams
  Padsevonil | 0.03914 (57.5) | 0.04054 (75.0) | 0.04987 (74.6)
  Metabolite 1 | 0.2101 (43.2) | 0.2333 (52.1) | 0.2309 (45.8)
  Metabolite 2 | 10.53 (42.5) | 9.423 (45.5) | 9.764 (53.1)
  Metabolite 3 | 29.11 (39.3) | 27.44 (42.3) | 26.09 (40.6)

22. Secondary Outcome: Cumulative Amount (Ae) of Padsevonil and Metabolites (1, 2, and 3) Excreted Into the Urine for Multiple Doses
Description: Ae: The cumulative amount of padsevonil and its metabolites (1, 2, and 3) excreted into the urine for multiple doses. Ae was expressed in milligrams (mg).
Time Frame: as for outcome 20
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 26
milligrams
  Padsevonil | 0.05825 (57.2) | 0.05741 (58.6) | 0.1274 (62.3)
  Metabolite 1 | 0.6188 (45.3) | 0.6657 (45.0) | 0.8797 (46.8)
  Metabolite 2 | 15.03 (45.8) | 15.07 (46.9) | 13.67 (41.4)
  Metabolite 3 | 70.83 (30.7) | 65.30 (34.0) | 81.36 (30.7)

23. Secondary Outcome: Fraction (fe) of Padsevonil and Metabolites (1, 2, and 3) Excreted Into the Urine for Single Dose
Description: fe: The fraction of padsevonil or metabolites (1, 2, and 3) excreted into the urine for single dose. fe was expressed in percentage (%).
Time Frame: Urine samples were taken 0 to 12 hours post first dose of Padsevonil during each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage excreted
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 27
percentage excreted
  Padsevonil | 0.03914 (57.5) | 0.04054 (75.0) | 0.04987 (74.6)
  Metabolite 1 | 0.2170 (43.2) | 0.2410 (52.1) | 0.2385 (45.8)
  Metabolite 2 | 10.52 (42.5) | 9.419 (45.5) | 9.760 (53.1)
  Metabolite 3 | 21.17 (39.3) | 19.96 (42.3) | 18.98 (40.6)

24. Secondary Outcome: Fraction (fe) of Padsevonil and Metabolites (1, 2, and 3) Excreted Into the Urine for Multiple Doses
Description: fe: The fraction of padsevonil and its metabolites (1, 2, and 3) excreted into the urine for multiple doses. fe was expressed in percentage (%).
Time Frame: as for outcome 20
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage excreted
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 26
percentage excreted
  Padsevonil | 0.05825 (57.2) | 0.05741 (58.6) | 0.1274 (62.3)
  Metabolite 1 | 0.6049 (45.6) | 0.6700 (44.6) | 0.8443 (45.3)
  Metabolite 2 | 15.02 (45.8) | 15.06 (46.9) | 13.15 (37.9)
  Metabolite 3 | 51.52 (30.7) | 47.50 (34.0) | 56.69 (38.0)

25. Secondary Outcome: Formation Clearance (CLform) of Padsevonil Metabolites (1, 2, and 3) in the Urine for Single Dose
Description: CLform: The formation clearance of padsevonil metabolites (1, 2, and 3) in the urine for single dose. CLform was expressed in milliliters per hour (mL/hour).
Time Frame: Urine samples were taken 0 to 12 hours post first dose of Padsevonil during each Treatment Period
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hour
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 27
mL/hour
  Metabolite 1 | 151.9 (67.3) | 153.4 (75.8) | 92.59 (80.8)
  Metabolite 2 | 7365 (80.2) | 5994 (87.8) | 3788 (107.5)
  Metabolite 3 | 14820 (60.5) | 12700 (59.9) | 7367 (72.0)

26. Secondary Outcome: Formation Clearance (CLform) of Padsevonil Metabolites (1, 2, and 3) in the Urine for Multiple Doses
Description: CLform: The formation clearance of padsevonil metabolites (1, 2, and 3) in the urine for multiple doses. CLform was expressed in milliliters per hour (mL/hour).
Time Frame: as for outcome 20
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/h
Arm/Group | Padsevonil (Period 1) (PK-PPS) | Padsevonil (Period 2) (PK-PPS) | Padsevonil and Erythromycin (Period 3b) (PK-PPS)
Number analyzed (Participants) | 28 | 28 | 26
mL/h
  Metabolite 1 | 295.3 (63.2) | 294.6 (58.9) | 166.4 (63.8)
  Metabolite 2 | 7331 (80.5) | 6622 (90.9) | 2593 (93.9)
  Metabolite 3 | 25150 (44.7) | 20890 (48.1) | 11170 (58.7)

27. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Serious Adverse Events (SAEs) During the Study
Description: An SAE is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Is an infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From beginning of the first Treatment Period (Day 1) to the Safety Follow-up Visit (up to 48 days )
Population: The Full Analysis Set (FAS) consisted of all study participants who have signed the Informed Consent form (ICF) and received investigational medicinal product (IMP). The analysis of this outcome measure was performed according to the treatment the participants actually received.
Measure: Number; unit: percentage of participants
Groups:
- Padsevonil (Period 1+2) (FAS): Treatment Period 1 (Day 1 to Day 11):
  * Padsevonil 100 mg bid on Day 1 to Day 4
  * Padsevonil 100 mg single dose on Day 5
  * 1 week of wash-out (from evening of Day 5 to Day 11)
  Treatment Period 2 (Day 12 to 22):
  * Padsevonil 100 mg bid on Day 12 to Day 15
  * Padsevonil 100 mg single dose on Day 16
  * 1 week of wash-out (from evening of Day 16 to Day 22). Study participants formed the Full Analysis Set (FAS).
- Erythromycin (Period 3a) (FAS): Study participants received Erythromycin in Treatment Period 3a as follows: 500 mg bid on Day 23 to Day 25. Study participants formed the FAS.
- Padsevonil and Erythromycin (Period 3b) (FAS): Study participants received Padsevonil and Erythromycin in Treatment Period 3b as follows:
  * Padsevonil 100 mg bid and erythromycin 500 mg bid on Day 26 to Day 32
  * Padsevonil 100 mg single dose on Day 33
  * Erythromycin 500 mg bid on Day 33. Study participants formed the FAS.
- Erythromycin (Period 3c) (FAS): Study participants received Erythromycin in Treatment Period 3c as follows: 500 mg bid on Day 34 to Day 37. Study participants formed the FAS.
Arm/Group | Padsevonil (Period 1+2) (FAS) | Erythromycin (Period 3a) (FAS) | Padsevonil and Erythromycin (Period 3b) (FAS) | Erythromycin (Period 3c) (FAS)
Number analyzed (Participants) | 28 | 27 | 27 | 26
percentage of participants | 0 | 0 | 0 | 0

28. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Non-serious Adverse Events (AEs) During the Study
Description: Treatment-emergent Adverse Events (TEAEs) were defined as those events which started on or after the date of first dose of UP0057 IMP, or events in which severity worsened on or after the date of first dose of UP0057 study medication.
Time Frame: From beginning of the first Treatment Period (Day 1) to the Safety Follow-up Visit (up to 48 days )
Population: The FAS consisted of all study participants who have signed the Informed Consent form ICF and received IMP. The analysis of this outcome measure was performed according to the treatment the participants actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Padsevonil (Period 1+2) (FAS) | Erythromycin (Period 3a) (FAS) | Padsevonil and Erythromycin (Period 3b) (FAS) | Erythromycin (Period 3c) (FAS)
Number analyzed (Participants) | 28 | 27 | 27 | 26
percentage of participants | 100 | 11.1 | 96.3 | 19.2

ADVERSE EVENTS:
Time Frame: From beginning of the first Treatment Period (Day 1) to the Safety Follow-up Visit (up to Day 48)
Description: FAS consisted of all study participants who have signed the ICF and received the IMP. The analysis was performed according to the treatment the participants actually received.
Arm/Group | Padsevonil (Period 1+2) (FAS) | Erythromycin (Period 3a) (FAS) | Padsevonil and Erythromycin (Period 3b) (FAS) | Erythromycin (Period 3c) (FAS)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27 | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 28/28 | 0/27 | 25/27 | 2/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Padsevonil (Period 1+2) (FAS) (N=28) | Erythromycin (Period 3a) (FAS) (N=27) | Padsevonil and Erythromycin (Period 3b) (FAS) (N=27) | Erythromycin (Period 3c) (FAS) (N=26)
Medical device site reaction (General disorders) | 5 (5) | 0 (0) | 7 (7) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 18 (27) | 0 (0) | 8 (8) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 28 (50) | 0 (0) | 25 (27) | 0 (0)
Depressed mood (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 6 (6) | 0 (0) | 5 (5) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT03480243/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT03480243/SAP_001.pdf